CLINICAL TRIAL: NCT03226353
Title: Performance of Somofilcon A Over One Week in Wearers Adapted to Omafilcon A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EX-MKTG-84
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Results first posted 2019-02-04 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- somofilcon A 1-day soft contact lenses (Experimental): Habitual and refitted wearers of omafilcon A were refit into somofilcon A for a week
  Interventions: Device: somofilcon A; Device: omafilcon A

INTERVENTIONS:
Device: somofilcon A — contact lens
Device: omafilcon A — contact lens

SUMMARY:
The objective of the study is to determine if habitual or adapted contact lens wearers of Omafilcon A can be confidently refit into Somofilcon A lenses and be successful after one week of daily wear.

The primary outcome variables for this study are:

* Investigator responses to refit questions;
* Lens fit.

DETAILED DESCRIPTION:
This is a prospective, single-site, dispensing, bilateral wear, open label, daily wear switch study, with the test lens (Somofilcon A) being worn for 7 (+5) days.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 17 years of age and has full legal capacity to volunteer;
* Has read and signed an information consent letter;
* Is willing and able to follow instructions and maintain the appointment schedule;
* Habitually wears soft spherical contact lenses with a power between +6.00 to -10.00D (inclusive) for a minimum 5 days per week, 10 hours per day and anticipates no difficulty wearing contact lenses for 7 days per week, 10 hours per day;
* Habitually wears, or is able to be adequately refit into Proclear 1 Day lenses;
* Demonstrates an acceptable fit with Proclear 1 Day and Clariti 1 Day contact lenses;
* Is correctable to a visual acuity of 0.20 LogMAR (approximately 20/30) or better (in each eye) with the study lenses or habitual correction;
* Manifest cylindrical spectacle refraction does not exceed -1.00DC in either eye.

Exclusion Criteria:

* Is participating in any concurrent clinical research study;
* Has any known active* ocular disease and/or infection;
* Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
* Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
* Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
* Is pregnant, lactating or planning a pregnancy at the time of enrolment (by verbal communication);
* Is aphakic;
* Has undergone refractive error surgery;
* Is an employee of the Centre for Contact Lens Research;
* Has taken part in another clinical or (pharmaceutical) research study within the last 7 days.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2017-09-27 (Actual); Study Completion 2017-09-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Participants: Habitual and refitted wearers of Omafilcon A were refitted with Somofilcon A
Period: Overall Study
Arm/Group | Overall Participants
Started | 77
Habitual Wearers of Proclear 1 Day | 2
Other Habitual Lens Types | 75
Completed | 71 (Study participants completed includes the Omafilcon A habitual wearers.)
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Screen Failure | 5

BASELINE CHARACTERISTICS:
Population: Two participants were habitual wearers of omafilcon A; the remaining participants were habitual wearers of other lens types. 71 subjects completed the study and 69 were included in analysis. One participant was excluded from all analysis due to protocol deviation and one participant was excluded from all analysis due to an adverse event.
Groups:
- Overall Participants: Habitual and refitted wearers of omafilcon A were refitted with somofilcon A. Two participants were habitual wearers of omafilcon A; the remaining participants were habitual wearers of other lens types. One participant was excluded from all analysis due to protocol deviation and one participant was excluded from all analysis due to an adverse event.
Arm/Group | Overall Participants
Number analyzed (Participants) | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 71
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 71

OUTCOME MEASURES:

1. Primary Outcome: Investigator Opinion On Overall Patient Refit From Omafilcon A to Somofilcon A: Does Somofilcon A Provides Easy and Quick Refit From Omafilcon A?
Description: Investigator level of agreement using a Likert scale on refitting participants from omafilcon A to somofilcon A at Visit 1 (Strongly Agree, Agree, Slightly Agree, Slightly Disagree, Disagree, Strongly Disagree)
Time Frame: 1 week
Population: Though 71 participants completed all protocol visits, two are completely excluded from all analyses. One participant was excluded because of three protocol deviations and other Participant was excluded because of an adverse event (non-significant ocular from Omafilcon A).
Measure: Count of Participants; unit: Participants
Groups:
- Overall Participants: Habitual and refitted wearers of Proclear 1 Day were refitted with Clariti 1 Day
Arm/Group | Overall Participants
Number analyzed (Participants) | 69
Participants
  Strongly disagree | 1
  Disagree | 0
  Slightly disagree | 13
  Slightly Agree | 11
  Agree | 32
  Styrongly agree | 12

2. Primary Outcome: Investigator Assessment to Refit- Based on the Investigator Opinion and Lens Fit Outcomes, Would the Investigator Refit the Subject Into Somofilcon A From Omafilcon A?
Description: Investigator level of agreement on the ease of refitting participants from omafilcon A to somofilcon A using Likert scale (Strongly agree, Agree, Slightly Agree, Slightly Disagree, Disagree, Strongly Disagree)
Time Frame: 1 week
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Participants
Number analyzed (Participants) | 69
Participants
  Strongly disagree | 0
  Disagree | 2
  Slightly disagree | 18
  Slightly agree | 20
  Agree | 18
  Strongly agree | 11

3. Primary Outcome: Investigator Assessment to Refit - Does Somofilcon A Performs Better Than Omafilcon A Day?
Description: as for outcome 2
Time Frame: 1 week
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Participants
Number analyzed (Participants) | 69
Participants
  Strongly disagree | 1
  Disagree | 3
  Slightly disagree | 30
  Sligtly agree | 19
  Agree | 14
  Strongly Agree | 2

4. Primary Outcome: Investigator Assessment to Refit - Does Somofilcon A Provides an Upgrade From Omafilcon A?
Description: as for outcome 2
Time Frame: 1 week
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Participants
Number analyzed (Participants) | 69
Participants
  Strongly Disagree | 1
  Disagree | 2
  Slightly Disagree | 19
  Slightly agree | 22
  Agree | 19
  Strongly agree | 6

5. Primary Outcome: Lens Fit - Post-blink Lens Movement
Description: Graded on a scale of 0-4, 1 step, 0=Insufficient, unacceptable movement, 4=Excessive, unacceptable movement.
Time Frame: Dispense and 1 Week
Population: 71 participants completed all protocol visits, two are completely excluded from all analyses because of protocol deviations and adverse event.Two participants were habitual wearers of omafilcon A lenses and not necessary to dispense new lenses.They are not included in the omafilcon A dispense analysis but included in the omafilcon A 1-week analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Somofilcon A; Omafilcon A: All participants that habitually wear omafilcon A and other contact lenses are refitted with omafilcon A for a week and then Fitted with somofilcon A for a week.
Arm/Group | Somofilcon A | Omafilcon A
Number analyzed (Participants) | 69 | 69
units on a scale
  Dispense: number analyzed (Participants) | 69 | 67
  Dispense | 2.1 (0.5) | 2.2 (0.5)
  1-week | 1.9 (0.6) | 2.0 (0.6)

6. Primary Outcome: Lens Fit - Lens Tightness
Description: Graded using 0-100 scale (5% steps) where 0 = extremely loose and 100 = extremely tight.
Time Frame: Dispense and 1 week
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Omafilcon A
Number analyzed (Participants) | 69 | 69
units on a scale
  Dispense: number analyzed (Participants) | 69 | 67
  Dispense | 48 (9) | 46 (7)
  1-week | 51 (8) | 47 (9)

7. Primary Outcome: Lens Fit - Lens Deposition
Description: Graded on a scale of 0-4, with 0.25 increments, 0=no deposits; 4=deposit ≥ 0.5mm or film >75% surface.
Time Frame: Dispense and 1 week
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Omafilcon A
Number analyzed (Participants) | 69 | 69
units on a scale
  Dispense: number analyzed (Participants) | 69 | 67
  Dispense | 0.38 (0.54) | 0.22 (0.33)
  1-week | 0.60 (0.63) | 0.36 (0.51)

8. Primary Outcome: Lens Fit - Centration
Description: (3 point scale: optimum, decentration acceptable, decentration unacceptable)
Time Frame: Dispense and 1 Week
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A | Omafilcon A
Number analyzed (Participants) | 69 | 69
Participants
  Dispense: number analyzed (Participants) | 69 | 67
  Dispense: Optimum | 26 | 40
  Dispense: Acceptable | 43 | 27
  Dispense: Unacceptable | 0 | 0
  1-week: Optimum | 28 | 35
  1-week: Acceptable | 41 | 34
  1-week: Unacceptable | 0 | 0

9. Primary Outcome: Lens Fit - Lens Wettability
Description: Graded on a scale of 0-4 with 0.25 increments, 0=excellent; 4=severely reduced.
Time Frame: Dispense and 1 Week
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Omafilcon A
Number analyzed (Participants) | 69 | 69
units on a scale
  Dispense: number analyzed (Participants) | 69 | 67
  Dispense | 0.54 (0.66) | 0.21 (0.34)
  1-week | 0.83 (0.78) | 0.42 (0.25)

10. Primary Outcome: Overall Lens Fit Acceptance
Description: Graded on a 0-4 point scale (where 0 = should not be worn, 4=perfect), providing a reason if Grade 2 or less
Time Frame: Dispense and 1 Week
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Omafilcon A
Number analyzed (Participants) | 69 | 69
units on a scale
  Dispense: number analyzed (Participants) | 69 | 67
  Dispense | 3.3 (0.6) | 3.6 (0.5)
  1-week | 3.2 (0.7) | 3.4 (0.7)

ADVERSE EVENTS:
Time Frame: From dispense to completion of follow up, approximately one week for each lens, two weeks total.
Groups:
- Somofilcon A; Omafilcon A: Habitual and refitted wearers of Proclear 1 Day were refitted with Clariti 1 Day. Two participants were habitual wearers of Proclear 1 day; the remaining were habitual wearers of other lens types.
Arm/Group | Somofilcon A | Omafilcon A
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/71
Other Adverse Events (participants affected / at risk) | 0/71 | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT03226353/Prot_SAP_001.pdf